CLINICAL TRIAL: NCT01349075
Title: A Humanitarian Device Exemption Treatment Protocol of Therasphere for the Treatment of Unresectable Hepatocellular Carcinoma
Brief Title: TheraSphere for the Treatment of Unresectable Hepatocellular Carcinoma
Status: Completed | Type: Observational
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Other Study IDs: 07D.366; 2007-49 (Other: CCRRC); JT 1283 (Other: JeffTrial Number)
Record Dates: First submitted 2011-05-04; First posted 2011-05-06 (Estimated); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Hepatocellular Carcinoma
Keywords: Unresectable; Hepatocellular Carcinoma; TheraSphere; Yttrium-90
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Yttrium-90

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- TheraSphere
  Interventions: Radiation: TheraSphere

INTERVENTIONS:
Radiation: TheraSphere — The target dose of TheraSphere most commonly used is 120 - 140 Gy. Standard radiation safety techniques will be used.
  Other Names: Yttrium-90

SUMMARY:
TheraSphere is a medical device containing yttrium-90 (Y-90) a radioactive material that has been used to treat liver tumors. When Y-90 is put into very tiny glass beads (TheraSphere), it can be injected into the liver through a blood vessel. This allows a large local dose of radiation to be delivered to the tumor with less risk of toxic effects from radiation to other parts of the body or to healthy liver tissue.

DETAILED DESCRIPTION:
Surgical resection of the affected portion of the liver offers the best chance for disease-free survival in patients with hepatoma (HCC). Unfortunately, most hepatoma patients present with disease that is not amenable to resection (multifocal disease) or have other medical contraindications to surgery (limited hepatic reserve related to advanced cirrhosis or chronic hepatitis). Fewer than 15%1 of hepatoma patients are suitable surgical candidates.

The objective of treatment with TheraSphere is to selectively administer a potentially lethal dose of radioactive material to neoplastic tissue in the liver of patients with HCC. Regional therapies for HCC may have several advantages over systemically administered treatments. Irradiating a cancer prior to treatment with regional chemotherapy may be more effective than either therapeutic modality alone. TheraSphere may also be of value as a 'bridging' treatment for HCC patients awaiting a donor organ for liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age, of any race or sex, who have hepatocellular carcinoma of the liver
* Patients who are able to give informed consent, will be eligible.
* Patients must have an ECOG Performance Status score of < or = 2
* Must have a life expectancy of > 3 months
* Non-pregnant with an acceptable contraception in premenopausal women
* Patients must be > 4 weeks since prior radiation or prior surgery and at least 1 month post chemotherapy

Exclusion Criteria:

* Contraindications to angiography and selective visceral catheterization
* Evidence of potential delivery of greater than 16.5 mCi (30 Gy absorbed dose) per treatment of radiation to the lungs
* Evidence of any detectable Tc-99m MAA flow to the stomach or duodenum, after application of established angiographic techniques to stop or mitigate such flow (ex. placing catheter distal to gastric vessels)
* Significant extrahepatic disease representing an imminent life-threatening outcome
* Severe liver dysfunction or pulmonary insufficiency
* Active uncontrolled infection
* Significant underlying medical or psychiatric illness
* Pregnancy
* Patients will be excluded if they have pre-existing diarrhea/illness, or if they have a co-morbid disease or condition that would preclude safe delivery of TheraSphere treatment and place the patient at undue risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from the patient population referred to the principal clinician for regional liver cancer therapy.
Sampling Method: Non-Probability Sample
Enrollment: 474 (Actual)
Dates: Start 2007-10; Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Response to Treatment | Through 24 months post-treatment
  Diagnostic imaging studies for assessment of tumor response will be performed according to usual standard of care as established by the referring oncologist. The principal clinician will be able to get a preliminary evaluation of tumor response in patients who return for subsequent treatment, as part of the imaging studies required for repeat safety screening of patients.

SECONDARY OUTCOMES:
Safety | Through 24 months post-treatment or death
  Evaluate toxicities and adverse experiences associated with TheraSphere treatment
Survival Time | Through 24 months post-treatment or death
  Evaluate survival time from the first treatment. The disease status, survival and safety status of all patients who receive TheraSphere treatment will be evaluated annually until death or 2 years post-treatment. In general, follow-up will be performed by the principal clinician. In the event of patient death, the date and cause of death will be recorded in the medical record (if possible).

CONTACTS AND LOCATIONS:
Overall Officials: Colette Shaw, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Kimmel Cancer Center at Thomas Jefferson University, an NCI-Designated Cancer Center — http://www.KimmelCancerCenter.org
- See also: Thomas Jefferson University Hospitals — http://www.JeffersonHospital.org/